CLINICAL TRIAL: NCT05973357
Title: The Influence of Vertical Implant Position With Immediate Provisionalization on the Marginal Bone Loss: A Randomized Controlled Clinical Trial
Brief Title: The Influence of Vertical Implant Position With Immediate Provisionalization on the Marginal Bone Loss.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, RWGWanis, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Dental Implant Failed; Implant Site Reaction
Keywords: Delayed Implant; Immediate loading; Temporization; provisionalization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-crestal group (Experimental): Patients receiving delayed implant placed 2mm sub-crestal level with immediate provisionalization
  Interventions: Procedure: Sub-crestal implant
- Equi-crestal grouo (Experimental): Patients receiving delayed implant placed equi-crestal level with immediate provisionalization
  Interventions: Procedure: Equi-crestal implant

INTERVENTIONS:
Procedure: Sub-crestal implant — Patients receiving delayed implant placed 2mm sub-crestal level with immediate provisionalization
  Arms: Sub-crestal group
Procedure: Equi-crestal implant — Patients receiving delayed implant placed equi-crestal level with immediate provisionalization
  Arms: Equi-crestal grouo

SUMMARY:
Multiple clinical studies have established high survival rates and tremendous predictability of dental implant treatment. However, a pleasant esthetic outcome is the patient's primary expectation regarding implants in the esthetic zone and several esthetic factors have been evaluated to contribute to an esthetic appearance. Among these, the midfacial soft tissue level is considered to be one of the most important factors; Cosyn and co-workers reported that among factors including soft tissue phenotype, the midfacial recession was associated with the position of the implant .

Therefore, subcrestal implant placement has been advocated as it has been associated with the reduction of crestal bone loss in cases with decreased soft tissue thickness. If the vertical soft tissues on the crest of the alveolar ridge are 2 mm or less at the time of implant placement, implants will undergo unavoidable bone resorption by establishing sufficient biologic protection. Another option was proposed by Linkevicius et al, who introduced the subcrestal implant placement as a method to accommodate the problem of thin soft tissues.

Research question:

Does the placement of delayed implants with different vertical depth affect the marginal bone loss with immediate provisionalization?

DETAILED DESCRIPTION:
Preservation of crestal bone is crucial and must be prioritized from the onset of implant placement. Adequate amount of peri-implant bone contributes to esthetic success and implant stability. Crestal bone contributes to both esthetics and function. Resorption of crestal bone is seen as loss of interproximal papillary support and gingival recession, which gives way to peri-implantitis and compromises esthetics.

With respect to the depth of insertion, implants can be placed at various levels in the bone, in which affects the peri-implant tissues with the surrounding marginal bone. Therefore, Placement of an implant in a deeper position with re¬spect to the bone crest (subcrestal placement) has been suggested as a method that could contribute to main¬tain the periimplant soft and hard tissues in comparison with crestal placement, though this affirmation is sub¬ject to controversy.

Rationale for conducting the research:

Limiting the extent of peri-implant bone loss has been recognized for decades to be an important aspect of long-term implant success, and stable peri-implant bone conditions play an important role in maintaining esthetics.

the opinion expressed widely in the scientific literature has been that subcrestal implant placement leads to increased crestal bone resorption. However, clinical studies addressing the implant placement depth in relation to crestal bone have been rare. Data on subcrestal versus crestal placement have mostly come from animal studies. Even fewer data are available regarding the effects of crestal versus subcrestal positioning of platform-switched implants.

In a prospective research, Nagarajan et al. implanted equicrestal and subcrestal implants to examine the crestal bone levels prior to loading. The crestal bone levels of the implants placed equicrestally (1.31 mm 1.04 mm and 0.68 mm 1.08 mm on mesial and distal surfaces, respectively) were higher than those of implants placed subcrestally (0.49 mm 0.49 mm and 0.025 mm 6.06 mm on mesial and distal surfaces, respectively), with a P value of crestal bone level for both groups being 0.12 and 0. They came to the conclusion that there was no difference in the amount of crestal bone loss prior to prosthetic loading between implants placed at subcrestal and equicrestal levels. In this study eqi-crestal implant will be used as a comparator but with immediate loading.

ELIGIBILITY:
Inclusion Criteria:

* ● Patients with single missing upper anterior or premolar teeth

  * Patients with minimum buccolingual width of 6 mm and mesiodistal width of 6mm
  * Patients with healthy systemic conditions.
  * Patients older than 18 years.
  * Good oral hygiene.
  * Accepts one year follow-up period (cooperative patients).
  * The patient provides informed consent.
  * Adequate Inter-arch space for implant placement.
  * Favorable occlusion (no traumatic occlusion).
  * Absence of allergy to the prescribed medications.

Exclusion Criteria:

* ● Patients with inadequate bone volume and/ or quality

  * Patients with local root remnants
  * Patients with inadequate wound healing
  * Patients with signs of acute infection related to the area of interest.
  * Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits (Lobbezoo et al., 2006).
  * Heavy smokers patients (more than 10 cigarettes per day) (Lambert, Morris and Ochi, 2000).
  * Metabolic diseases such as diabetes or hyperthyroidism as well as systemic medications such as chemotherapy or bisphosphonates
  * Pregnant or nursing women.
  * Uncooperative patients.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss | 1 year follow up
  Crestal bone loss

SECONDARY OUTCOMES:
Mid facial recession | 1 year follow up
  Corono-apical distance between the peri-implant soft tissue margin and the cemento-enamel junction (CEJ) of the homologous contralateral tooth. Midfacial recession will be measured at 6, and 12 months.
The pink esthetic score | 1 year follow up
  The pink esthetic score will be calculated on the parameters defined by. Clinical photographs will be taken to evaluate peri-implant soft tissue through evaluating seven variables compared to a natural reference tooth including: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value. The maximum achievable PES is 14.
Gingival Thickness | 1 year follow up
  Gingival thickness will be measured using an anesthetic needle with a rubber stopper, trans-gingivally piercing tissues horizontally perpendicular to the long axis of the tooth/implant until it contacts bone, at 3 different points; three readings mid-buccally at three different levels; 2mm, 4mm and 6mm apical to the gingival margin. The length of the part of the instrument that penetrates into the soft tissue is measured in mm using a digital caliper (Wiesner et al., 2010).
Implant Survival | 1 year follow up
  A binary outcome, the definition of implant success was based on the clinical and radiographic criteria;1) absence of clinically detectable implant mobility; 2) absence of pain or any subjective sensation; 3) absence of recurrent peri-implant infection; and 4) absence of persistent radiolucency around the implant after 12 months of loading
Post-operative patient satisfaction | 1 year follow up
  A 12-items questionnaire are self-reported by the patients after 12 months post-operative; 6 questions with with visual analoge scale from 1 to 10 with poorest score is not very satisfied equal 0 and optimum score is satisfied which equals 10. The another 6 questions is yes or no questions
  This questions measure patient's acceptability and esthetics satisfaction

IPD SHARING:
Plan to Share IPD: Undecided